CLINICAL TRIAL: NCT01126801
Title: Effects of Estrogen and Hot Flashes on Mood in Postmenopausal Women
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Stopped enrolling subjects due to challenge of identifying eligible participants
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Hadine Joffe, MD, Vice Chair for Research, Psychiatry Department, Brigham and Women's Hospital
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2009p001776
Record Dates: First submitted 2010-05-11; First posted 2010-05-20 (Estimated); Results first posted 2016-08-22 (Estimated); Last update posted 2017-10-20 (Actual); Status verified 2017-09

CONDITIONS: Menopausal Depression
MeSH Terms: interventions — Estradiol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Estradiol (Experimental)
  Interventions: Drug: Estradiol
- Placebo control (Placebo Comparator)
  Interventions: Other: Placebo control

INTERVENTIONS:
Drug: Estradiol — Oral estradiol 1.0 mg/day for four weeks.
  Arms: Estradiol
Other: Placebo control — Placebo control matched to estradiol tablets. Daily dosing for one month.
  Arms: Placebo control

SUMMARY:
This protocol is a controlled study of estradiol therapy in early postmenopausal women with and without frequent hot flashes that will be used to determine whether hot flashes are an important intermediary in the generation of menopause-associated depression.

DETAILED DESCRIPTION:
SPECIFIC AIMS (Research Objectives)

To define the relative effects of hot flashes and changes in estradiol on mood in postmenopausal women:

Hypotheses:

1. Estrogen treatment has a similar therapeutic effect on mood in women with and without frequent hot flashes
2. Estradiol levels correlate with improvement in mood

ELIGIBILITY:
Inclusion Criteria:

* Healthy women ≥40 years-old
* Early postmenopausal, defined as:
* No menstrual bleeding for 12-60 months secondary to natural menopause, according to STRAW criteria48
* Hysterectomy without bilateral oophorectomy if surgery was completed after 6+ months of amenorrhea (no maximum duration of amenorrhea required)
* Bilateral oophorectomy (no minimum or maximum duration of amenorrhea required)
* Serum follicle-stimulating hormone (FSH) >25 IU/L and estradiol <20 pg/ml
* Diagnosis of major depression on the MINI
* Mild-to-moderate depressive symptoms, as indicated by MADRS score 15-31 and BDI score >15
* Normal mammogram within the past 2 years
* Good general health

Exclusion Criteria:

* Severe depression, defined as a MADRS score >31, psychotic symptoms, or suicidal or homicidal ideation
* Psychiatric illness, as defined by clinical interview and the Mini-International Neuropsychiatric Interview (MINI), as:

  * A lifetime history of bipolar disorder
  * A lifetime history of severe depression, as characterized by current or prior psychotic symptoms, inpatient psychiatric hospitalization or a suicide attempt in the previous 5 years, or
  * Current panic disorder or obsessive compulsive disorder
  * A lifetime history of psychotic symptoms
  * Current anorexia nervosa
  * An alcohol or substance-use disorder active within the past year
  * Current suicidal or homicidal ideation
* Previous diagnosis of a sleep disorder (sleep apnea, PLMS, etc) or diagnosed on a screening PSG study
* Pregnant, confirmed with serum ß-HCG at baseline (Visit 1)
* Breastfeeding
* Contraindication, hypersensitivity, or previous adverse reaction to E2 therapy
* Current or recent (1 month) use of centrally active medications (antidepressants, anxiolytics, hypnotics, anticonvulsants, stimulants)
* Current or recent (2 months) use of systemic hormone medications
* History of breast cancer, premalignant breast lesions, or undiagnosed breast mass
* Vaginal spotting or bleeding
* History of thrombo-embolism, cardiovascular disease, congestive heart failure or other contraindication to estradiol therapy.
* Liver dysfunction or disease
* Renal insufficiency
* Contraindications to progestin therapy
* Asthma, diabetes mellitus, epilepsy, and migraine disorders that are not stable and under medical management
* Other medical contraindications to estradiol and progestin therapy including porphyria, systemic lupus erythematosus, hepatic hemangiomas, deep vein thrombosis, hereditary angioedema, hypertriglyceridemia, severe Hypocalcemia.
* Clinically significant abnormalities in screening blood tests including:

  * Thyroid-stimulating hormone <0.50 or >5.0 uU/mL)
  * Shift workers

Min Age: 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2010-05; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hadine Joffe, MD MSc, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Galvan T, Camuso J, Sullivan K, Kim S, White D, Redline S, Joffe H. Association of estradiol with sleep apnea in depressed perimenopausal and postmenopausal women: a preliminary study. Menopause. 2017 Jan;24(1):112-117. doi: 10.1097/GME.0000000000000737. PMID 27648659

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo control: Placebo control matched to estradiol tablets. Daily dosing for one month.
Period: Overall Study
Arm/Group | Estradiol | Placebo
Started | 1 | 1
Completed | 1 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Estradiol | Placebo | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 50 (0) | 55 (0) | 52.5 (3.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Improvement of Mood, Measured by the Clinician-rated Montgomery-Asberg Depression Rating Scale (MADRS) From Baseline to Study End.
Time Frame: one month
Population: No participants were analyzed since the study was terminated due to difficulty recruiting subjects. Because data from only one subject per arm were collected, these data are not reported to preserve subject privacy.
Arm/Group | Estradiol | Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Improvement of Mood, Measured by the Self-rated Beck Depression Inventory (BDI) From Baseline to Study End.
Time Frame: one month
Population: as for outcome 1
Arm/Group | Estradiol | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Estradiol | Placebo
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 0/1 | 0/1

LIMITATIONS AND CAVEATS:
Due to the challenge of identifying eligible participants, we decided to stop enrolling subjects and not to analyze the 2 completed participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No